CLINICAL TRIAL: NCT00885612
Title: 10-year CHD Risk Evaluation and Its Treatment Pattern Analysis in Postmenopausal Early Breast Cancer Patients Taking Aromatase Inhibitors
Brief Title: 10 Year Coronary Heart Disease (CHD) Risk Evaluation and Its Treatment Pattern Analysis in Postmenopausal Early Breast Cancer (EBC) Patients Taking Aromatase Inhibitors (AI)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-OKR-DUM-2009/1
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer
Keywords: CHD-Risk; Breast Cancer; Aromatase Inhibitors; postmenopausal early breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
10-year CHD risk evaluation and its treatment pattern analysis in postmenopausal early breast cancer patients taking aromatase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Early Breast Cancer patients
* Postmenopausal Status
* patients taking Aromatase Inhibitor as adjuvant treatment no longer than 6 months

Exclusion Criteria:

* Advanced Breast Cancer patients(stage iii, iv)
* Patients who are hard to be analysed by limitation of chart record according to investigators discretion
* patients who already have been registered in this study

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal patients with early breast cancer, who are taking aromatase inhibitors no longer than 6 months as an adjuvant treatment after surgery
Sampling Method: Probability Sample
Enrollment: 1114 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to define 10-year CHD risk according to Framingham risk score in postmenopausal early breast cancer patients who are taking aromatase inhibitors as an adjuvant treatment. | 1 visit

SECONDARY OUTCOMES:
To describe 10-year CHD risk comparing to the historical data of 10-year cancer-specific mortality in breast cancer | 1 Visit
To analyse CHD management patterns according to defined 10-year CHD risk categories | 1 Visit
To describe correlation between concommitant medication(Anthracycline, Trasuzumab) and CHD risk | 1 Visit

CONTACTS AND LOCATIONS:
Overall Officials: JoonWoo Bahn, MD, PhD, Study Director — AstraZeneca Korea
Locations (27):
- South Korea (27):
  - Research Site, Cheonan, Chungcheongnam-do
  - Research Site, Chuncheon, Gangwon-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Pohang, Gyeongsangbuk-do
  - Research Site, Masan-si, Gyeongsangnam-do
  - Research Site, Anyang
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gangneung
  - Research Site, GuangJu
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Inchon
  - Research Site, Jeonju
  - Research Site, Junam
  - Research Site, Koyang
  - Research Site, Kyunggi
  - Research Site, Pusan
  - Research Site, Seoul
  - Research Site, Seoul(Kangbuk)
  - Research Site, Seoul(Kangdong)
  - Research Site, Seoul(Kangnam)
  - Research Site, Seoul(Yeouido)
  - Research Site, Suwon
  - Research Site, Ulsan